CLINICAL TRIAL: NCT03981237
Title: Postoperative Pain After Ultrasonically and Laser-activated Irrigation During Root Canal Treatment: a Randomized Clinical Trial
Brief Title: Postoperative Pain After Ultrasonically and Laser-activated Irrigation During Root Canal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B670201939441
Record Dates: First submitted 2019-05-27; First posted 2019-06-10 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2020-04

CONDITIONS: Post-operative Pain
Keywords: root canal treatment; root canal irrigation
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Root canal treatment with laser-activated irrigation (Experimental): In these patients, the root canals of the tooth are chemomechanically prepared. After shaping, irrigant activation is performed by means of a pulsed erbium laser. The canals are then dried and obturated.
  Interventions: Device: Laser-activated irrigation with a pulsed Er:YAG laser; Procedure: Orthograde root canal treatment
- Root canal treatment with ultrasonically activated irrigation (Active Comparator): In these patients, the root canals of the tooth are chemomechanically prepared. After shaping, irrigant activation is performed by means of an ultrasonically driven instrument. The canals are then dried and obturated.
  Interventions: Device: Ultrasonically activated irrigation; Procedure: Orthograde root canal treatment

INTERVENTIONS:
Device: Laser-activated irrigation with a pulsed Er:YAG laser — The root canals and the pulp chamber are filled with NaOCl 3%. Per canal, the laser tip is placed above the root canal entrance and activated (frequency 20 Hz, pulse energy 20 mJ and pulse length 50 μs) for 30s. TThe canal is then rinsed with NaOCl using a 27G needle, followed by a second application of laser, identical to the first.
  Arms: Root canal treatment with laser-activated irrigation
Device: Ultrasonically activated irrigation — The root canals and the pulp chamber are filled with NaOCl 3%. An Irrisafe file, driven by an ultrasonic unit according to the manufacturers' instructions, is held at 1-3 mm from WL (precurved if canal is curved) and activated for 30 s. The canal is then rinsed with NaOCl using a 27G needle. This cycle is repeated three times (i.e. 3*20s).
  Arms: Root canal treatment with ultrasonically activated irrigation
Procedure: Orthograde root canal treatment — After rubber dam isolation and field disinfection, the pulp chamber is accessed. The root canal(s) is/are located and shaped using manual and mechanical NiTi instruments in combination with NaOCl (3%) irrigant. The canals are dried using paper points and obturated with gutta percha and epoxy resin sealer. The tooth is sealed with a temporary or permanent filling.

SUMMARY:
The aim of this prospective, randomized clinical study is to compare the frequency and intensity of post-operative pain after root canal treatment with ultrasonically-activated or laser-activated irrigation.

DETAILED DESCRIPTION:
Patients older than 18 years who require root canal treatment of an asymptomatic tooth with vital or necrotic pulp are included. Those teeth are subjected to root canal treatment using hand and rotating/reciprocating instruments, in combination with irrigation (3% NaOCl, 17% EDTA). After chemomechanical preparation, the teeth are randomly allocated to one of the following groups, according to the final irrigant activation:

* Ultrasonically activated irrigation (UAI), with an Irrisafe file (Satelec Acteon, Mérignac, France) held 1-3mm from working length, driven by an ultrasonic device, activated for 3 x 20 seconds. In between each 20-second cycle, each canal is rinsed with 1 mL NaOCl and finally with 2 mL.
* Laser-activated irrigation (LAI), with the tip of a pulsed Er:YAG laser (2940 nm, Fidelis II, Fotona) held above the canal entrance, activated for 2 x 30s. Settings are 20 Hz, 50 μs, 20 mJ. In between each 30-second cycle, each canal is rinsed with 1 mL NaOCl and finally with 2 mL.

The canals are then dried using paper points and obturated with gutta percha and an epoxy resin sealer using warm vertical condensation. Finally, the endodontic access is sealed with a provisional or permanent filling.

The patient is asked to keep a pain diary after the treatment, indicating postoperative pain on a visual analogue scale at 6, 24, 48 and 72 hours after treatment. Pain medication (Ibuprofen 400mg) is prescribed, and the intake of analgesic tablet is recorded at the same times.

Pre-Treatment Procedure

* Medical + dental history
* Clinical examination: sensibility tests, percussion, palpation, mobility, pockets measurement
* Radiographic examination
* Pulpal and periapical diagnosis
* Intensity of pre-op pain on 100mm VAS scale
* Patient information and informed consent
* Explanation on how to complete the pain diary and how and when to return it

Endodontic Protocol

* Anesthesia
* Rubber dam, disinfection of operative field
* Removal of caries and/or defective restorations
* Access cavity
* Build-up to provide a reservoir for the irrigation if necessary
* Crown-down preparation
* Length determination
* Apical enlargement

Irrigation protocol

* 3% NaOCl
* 17% EDTA when shaping completed
* Irrigation throughout the whole procedure with 27G notched-end needle 2 - 3 mm from WL

ELIGIBILITY:
Inclusion Criteria:

* subject has an asymptomatic (VAS 0-0,4mm) tooth requiring primary endodontic treatment
* subject must be able to undergo primary endodontic treatment

Exclusion Criteria:

* analgesic intake over the last 12h
* immunocompromised patients
* pregnant women
* tooth with incompletely formed apex/apices
* subjects with more than one tooth in need of RCT
* previously root canal treated teeth
* subjects with intolerance on NSAID's

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Level of post-operative pain after 24 hours | 24 hours after intervention
  Self-reported pain intensity at 24h after intervention, indicated on a 100mm Visual Analogue Scale. The VAS is a straight line with one end (point 0) meaning no pain and the other end( point 10) meaning the worst pain imaginable.
Level of post-operative pain after 6 hours | 6 hours after intervention
  Self-reported pain intensity at 6h after intervention, indicated on a 100mm Visual Analogue Scale. The VAS is a straight line with one end (point 0) meaning no pain and the other end( point 10) meaning the worst pain imaginable.
Level of post-operative pain after 48 hours | 48 hours after intervention
  Self-reported pain intensity at 48h after intervention, indicated on a 100mm Visual Analogue Scale. The VAS is a straight line with one end (point 0) meaning no pain and the other end( point 10) meaning the worst pain imaginable.
Level of post-operative pain after 72 hours | 72 hours after intervention
  Self-reported pain intensity at 72h after intervention, indicated on a 100mm Visual Analogue Scale. The VAS is a straight line with one end (point 0) meaning no pain and the other end( point 10) meaning the worst pain imaginable.

SECONDARY OUTCOMES:
Analgesic intake | 6, 24, 48, 72 hours after intervention
  Number of analgesic tablets (Ibuprofen 400mg) taken at 6, 24, 48 and 72h after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Ziekenhuis Gent, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liapis D, De Bruyne MAA, De Moor RJG, Meire MA. Postoperative pain after ultrasonically and laser-activated irrigation during root canal treatment: a randomized clinical trial. Int Endod J. 2021 Jul;54(7):1037-1050. doi: 10.1111/iej.13500. Epub 2021 Mar 9. PMID 33595920